CLINICAL TRIAL: NCT04059250
Title: Nobio In Situ Clinical Study - Pilot Study
Brief Title: Nobio Clinical Study - Demineralization Prevention With a New Antibacterial Restorative Composite
Acronym: Nobio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Nobio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P0535966
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Results first posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries; Denture, Partial, Removable
Keywords: composite bactericidal; caries prevention
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: In-situ testing using a gap model inside the two flanges of a removable partial denture
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects are not aware, which side of the denture will harbor the gap model with the Nobio composite and which side harbors the traditional composite.
  Laboratory microhardness measurements will be conducted while keeping the operator blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Nobio flange (Experimental): On the Nobio flange side of the lower partial denture the gap model will include a double sterilized piece of human enamel, a small gap, and next to it the Nobio composite.
  Interventions: Device: Nobio composite
- Traditional composite flange (Placebo Comparator): On the traditional composite flange side of the lower partial denture the gap model will include a double sterilized piece of human enamel, a small gap, and next to it a traditional composite.
  Interventions: Device: traditional composite

INTERVENTIONS:
Device: Nobio composite — Nobio has developed a bactericidal composite, which does not leak out the bactericidal nano fillers
  Arms: Nobio flange
Device: traditional composite — traditional composite which has no bactericidal activities
  Arms: Traditional composite flange

SUMMARY:
Nobio has developed dental restorative materials with long term antibacterial properties in order to fight recurrent decay/caries around restorations. These composites with incorporated non-leaching antibacterial agents might overcome the vicious circle of newly developed cavities around freshly placed fillings.

The investigators will ask lower partial denture wearers to allow them to place a "gap model" with the Nobio-composite and enamel slab in one denture flange. In the other denture flange a gap model with a standard composite will be placed as control. In the laboratory the investigators will test with established methods for demineralization/caries prevention in the test and control enamel slabs, respectively.

DETAILED DESCRIPTION:
As a major issue in dentistry, it has been stated that two-thirds of all restorative dentistry involves the replacement of failed restorations. Secondary caries indicates a lesion developing at the margins of an existing restoration and is the major reason for replacement of amalgam and composite resin restorations in operative dentistry.

In research the use of experimental intra-oral caries models dealing with caries prevention has increased. The most realistic experimental model is the in vivo model that uses living teeth, followed by the in situ model using specimens with natural surfaces held in the mouth during the experimental period. In situ models have the potential to study both fundamental aspects of the caries process as well as more applied research problems in caries prevention in human subjects without actually causing caries in the natural dentition.

To simulate a failed interface between a tooth and a restoration, a gap can be formed between an enamel slab and the restoration prior to a cariogenic challenge. The "gap-model" will be inserted for instance into the denture flanges, and the cariogenic challenge occurs inside the mouth during the wear period..

Nobio has developed dental restorative materials with long term antibacterial properties in order to fight recurrent decay around restorations. These composites with incorporated non-leaching antibacterial agents might overcome the vicious circle of newly developed cavities around freshly placed fillings. The ongoing caries activity due to bacteria around the filling may be interrupted by quaternary ammonium silica dioxide (QASi) particles incorporated in the test composite at 1.2% (by weight). These particles are members of the Nobio Antimicrobial Particle (NAP) family (Nobio, Israel). QASi are synthesized to form a high concentration of antimicrobial groups that are covalently-bound onto a carrier core, such as silica. The resulting micro or nano-sized QASi particles are mixed with other fillers of the dental composite material, during manufacturing. Following in situ placement and light-initiated polymerization, QASi particles are permanently retained in the final dental restoration. Laboratory studies have shown that the quaternary ammonium silica particles are potent antibacterial agents, do not leach out in contrast to other antimicrobials or caries preventive active substances, inhibit the breakdown of the composite, and maintain antibacterial activity over time.

The study is an in situ study. Subjects, wearing lower partial dentures with acrylic flanges on both sides of the mouth will be recruited. On each side of the denture an enamel slab will be placed next to a composite, separated by a tiny gap. On one side of the denture the composite will be Nobio's antibacterial composite, on the other side a regular composite (a Nobio composite w/o particles or another commercial composite will serve as control material. Enamel slab and composite will be recessed into the flange, allowing microbial plaque to accumulate on top of it and especially in the gap.

After wearing the dentures for four weeks with the slabs, decalcification - ΔZ mineral loss - in the enamel slabs adjacent to the gap will be determined by cross-section microhardness testing in the laboratory. Average ΔZ mineral loss will be calculated for the Nobio group and the control group, and difference will be tested for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80 years,
* have at least six natural teeth remaining and have a recent history of dental caries
* wearing lower partial denture (with replaced teeth on both sides of the mouth)
* willing to wear their denture during the night
* are in good health, of either gender
* are in good current oral health with no active caries or periodontal disease (but with a history of caries)
* have an understanding of the study
* have saliva flow within the normal range (stimulated saliva flow rate of greater than 0.7 ml/minute)
* no antibiotics for the last three months
* willing to comply with all study procedures and protocols,
* residing in San Francisco or other nearby locales with community water fluoridation (to eliminate water fluoridation as a potential confounding variable)
* able to give written consent themselves
* must be able to read and understand English
* willing to sign the "Authorization for Release of Personal Health Information and Use of Personally Unidentified Study Data for Research" form; data will only be used for research

Exclusion Criteria:

* subjects who have less than 6 natural teeth remaining
* subjects who have used a 5,000 ppm fluoride toothpaste in the last 6 months
* subjects who have used Chlorhexidine or any other antimicrobials (cetylpyridinium etc.) in the last 6 months
* show evidence of extremely poor oral hygiene
* subjects suffering from systemic diseases, significant past or medical history with conditions that may affect oral health or oral flora (i.e. diabetes, HIV, heart conditions that require antibiotic prophylaxis)
* taking medications that may affect the oral flora or salivary flow (e.g. antibiotic use in the past three months, drugs associated with dry mouth / xerostomia)
* other conditions that may decrease the likelihood of adhering to study protocol
* in-office fluoride treatment within the last three months
* subjects who will leave the area and are unable to complete the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rechmann, Principal Investigator — UCSF - School of Dentistry - Preventive and Restorative Dental Sciences
Locations (1):
- UCSF School of Dentistry, Preventive and Restorative Dental Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clasen AB, Ogaard B. Experimental intra-oral caries models in fluoride research. Acta Odontol Scand. 1999 Dec;57(6):334-41. doi: 10.1080/000163599428580. PMID 10777137
- [Background] Zero DT. In situ caries models. Adv Dent Res. 1995 Nov;9(3):214-30; discussion 231-4. doi: 10.1177/08959374950090030501. PMID 8615944
- [Background] Gorton J, Featherstone JD. In vivo inhibition of demineralization around orthodontic brackets. Am J Orthod Dentofacial Orthop. 2003 Jan;123(1):10-4. doi: 10.1067/mod.2003.47. PMID 12532056
- [Background] Maupome G, Sheiham A. Criteria for restoration replacement and restoration life-span estimates in an educational environment. J Oral Rehabil. 1998 Dec;25(12):896-901. doi: 10.1046/j.1365-2842.1998.00328.x. PMID 9888223
- [Background] Kidd EA. Diagnosis of secondary caries. J Dent Educ. 2001 Oct;65(10):997-1000. PMID 11700003
- [Background] Hals E, Nernaes A. Histopathology of in vitro caries developing around silver amalgam fillings. Caries Res. 1971;5(1):58-77. doi: 10.1159/000259733. No abstract available. PMID 5277150
- [Background] Kuper NK, Montagner AF, van de Sande FH, Bronkhorst EM, Opdam NJ, Huysmans MC. Secondary Caries Development in in situ Gaps next to Composite and Amalgam. Caries Res. 2015;49(5):557-63. doi: 10.1159/000438728. Epub 2015 Sep 26. PMID 26407050
- [Background] Hollanders ACC, Kuper NK, Maske TT, Huysmans MDNJM. Secondary Caries in situ Models: A Systematic Review. Caries Res. 2018;52(6):454-462. doi: 10.1159/000487200. Epub 2018 Apr 5. PMID 29621757
- [Background] Benelli EM, Serra MC, Rodrigues AL Jr, Cury JA. In situ anticariogenic potential of glass ionomer cement. Caries Res. 1993;27(4):280-4. doi: 10.1159/000261551. PMID 8402802
- [Background] Dijkman GE, Arends J. Secondary caries in situ around fluoride-releasing light-curing composites: a quantitative model investigation on four materials with a fluoride content between 0 and 26 vol%. Caries Res. 1992;26(5):351-7. doi: 10.1159/000261467. PMID 1468099
- [Background] Beyth N, Yudovin-Farber I, Bahir R, Domb AJ, Weiss EI. Antibacterial activity of dental composites containing quaternary ammonium polyethylenimine nanoparticles against Streptococcus mutans. Biomaterials. 2006 Jul;27(21):3995-4002. doi: 10.1016/j.biomaterials.2006.03.003. Epub 2006 Mar 27. PMID 16564083
- [Background] Beyth N, Houri-Haddad Y, Baraness-Hadar L, Yudovin-Farber I, Domb AJ, Weiss EI. Surface antimicrobial activity and biocompatibility of incorporated polyethylenimine nanoparticles. Biomaterials. 2008 Nov;29(31):4157-63. doi: 10.1016/j.biomaterials.2008.07.003. Epub 2008 Aug 3. PMID 18678404
- [Background] Beyth N, Yudovin-Fearber I, Domb AJ, Weiss EI. Long-term antibacterial surface properties of composite resin incorporating polyethyleneimine nanoparticles. Quintessence Int. 2010 Nov-Dec;41(10):827-35. PMID 20927419
- [Background] Chatzistavrou X, Velamakanni S, DiRenzo K, Lefkelidou A, Fenno JC, Kasuga T, Boccaccini AR, Papagerakis P. Designing dental composites with bioactive and bactericidal properties. Mater Sci Eng C Mater Biol Appl. 2015;52:267-72. doi: 10.1016/j.msec.2015.03.062. Epub 2015 Mar 28. PMID 25953567
- [Derived] Rechmann P, Le CQ, Chaffee BW, Rechmann BMT. Demineralization prevention with a new antibacterial restorative composite containing QASi nanoparticles: an in situ study. Clin Oral Investig. 2021 Sep;25(9):5293-5305. doi: 10.1007/s00784-021-03837-4. Epub 2021 Feb 19. PMID 33608748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: each participant enrolled had TWO flanges (right and left side of the mouth) in her/his removable partial denture; the study design is a split-mouth design - in one side the "Nobio Flange"- the Nobio composite was inserted, one the control side - the "control flange" - the traditional control composite was inserted
Units Other Than Participants: right or left flange of one denture
Groups:
- Traditional Composite Control Flange: On the traditional control composite flange side of the lower partial denture the gap model will include a double sterilized piece of human enamel, a small gap, and next to it a traditional control composite.
  traditional composite: traditional composite which has no bactericidal activities
Period: Overall Study
Arm/Group | Nobio Flange | Traditional Composite Control Flange
Started | 25; 25 right or left flange of one denture | 25; 25 right or left flange of one denture
Completed | 25; 25 right or left flange of one denture | 25; 25 right or left flange of one denture
Not Completed | 0; 0 right or left flange of one denture | 0; 0 right or left flange of one denture

BASELINE CHARACTERISTICS:
Population: 25 participants contributed 25 lower partial dentures. Each partial denture had two flanges - one side for the Nobio unit, the other side as the control composite unit
Groups:
- All Study Participants: All participants received both the Nobio flange and the traditional composite control flange.
  On the Nobio flange side of the lower partial denture the gap model will include a double sterilized piece of human enamel, a small gap, and next to it the Nobio composite.
  Nobio composite: Nobio has developed a bactericidal composite, which does not leak out the bactericidal nano fillers
  On the traditional composite control flange side of the lower same partial denture the gap model will include a double sterilized piece of human enamel, a small gap, and next to it a traditional composite.
  traditional composite: traditional composite which has no bactericidal activities
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Mineral Loss ΔZ
Description: The mineral loss is determined in the laboratory using cross-sectional microhardness testings of the enamel after the 4-weeks wearing period of the gap-model.
  The overall relative mineral loss, ΔZ, for each sample is calculated by creating a hardness profile curve by plotting normalized volume percent mineral against distance from the outer enamel surface. The area under the curve that represents ΔZ (µm * vol % mineral) is calculated using Simpson's integration rule.
Time Frame: mineral loss ΔZ is determined after the 4 week wearing period
Population: From the original 25 subjects data of the first 5 subjects were used for a sample size calculation. The sample size calculation determined data from 17 subjects would be needed. To account for loss due to follow-up issues, we recruited 20 subjects. 1 subject did not follow the instructions (required wearing time), 2 sample/data sets could not be retrieved due to Covid-19 shelter-in-place restrictions. Results of the first 5 were not included due to statisticians concerns for clean statistics.
Measure: Mean (Standard Deviation); unit: vol% * μm]
Arm/Group | Nobio Flange | Traditional Composite Flange
Number analyzed (Participants) | 17 | 17
vol% * μm] | 235 (354) | 774 (556)

ADVERSE EVENTS:
Time Frame: Four weeks study period, while wearing the composite inside the denture flanges
Arm/Group | Nobio Flange | Traditional Composite Flange
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT04059250/Prot_SAP_001.pdf